CLINICAL TRIAL: NCT07162532
Title: Impact of Clinico-hematological and Molecular Characteristics on Treatment Outcomes of Chronic Lymphocytic Leukemia Patients
Brief Title: Clinico-hematological and Molecular Characteristics of Chronic Lymphocytic Leukemia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, sawsan abdelllah, specialist of clinical hematology, Assiut University
Other Study IDs: molecular characters of CLL
Record Dates: First submitted 2025-07-11; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

INTERVENTIONS:
Diagnostic Test: 1 Complete blood picture (CBC) with blood film, lymphocytic count 2 and viral hepatitis 3 Immunophenotyping 4 LDH 5 Coomb's tests ,deletion 17p,IGVH mutation,ESR — Complete blood picture (CBC) with blood film, lymphocytic count 2 Routine liver and kidney function and viral hepatitis 3 Immunophenotyping 4 LDH 5 Coomb's tests 6 Erythrocyte sedimentation rate (ESR). 7 C reactive protein (CRP). 8 Cytogenetic profiles: del(17p) 9 molecular study :IGHV mutation status.

SUMMARY:
the goal of this study is To describe the clinical, hematologic, and cytogenetic characteristics of CLL cases.

The main questions it aims to answer are:

1. what is the impact of cytogenetics abnormalities [e.g., IGHV mutation status, del(17p)] on patients' treatment response?
2. what is th correlation between clinical and hematological characteristic with patients' outcome.

All participants will be subjected to history taking , Physical examination. and Laboratory investigations (Complete blood picture Cytogenetic profiles: del(17p) molecular study :IGHV mutation status).

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukemia (CLL) is a CD 5 positive hematological malignancy that is characterized by the excess accumulation of small, mature appearing neoplastic B lymphocytes in the blood, marrow, and other lymphoid tissues, resulting in lymphocytosis, leukemia cell infiltration of the marrow, lymphadenopathy, and splenomegaly. Clonal B lymphocytes with a distinctive immunophenotype where B-cell markers (CD19, CD23) are expressed along with CD5, with low-level expression of CD20 and surface immunoglobulins . CLL is more common in men than women, and its incidence varies geographically, with higher rates reported in Western countries [5]. Clinical characteristics in the form of organomegaly and lymphadenopathy in addition to hematological characteristics in the form of lymphocytosis and cytopenia affect disease coarse and patients' outcome .The clinical course of CLL is highly variable, ranging from indolent disease that may never require treatment to aggressive forms that necessitate prompt intervention. Some patients may remain asymptomatic for many years, while others may experience symptoms such as fatigue, weight loss, and recurrent infections due to immune dysfunction . Cytogenetic and molecular genetic studies have identified a range of genetic abnormalities in CLL, including deletions, translocations, and mutations . These genetic alterations can affect the behavior of the disease and influence treatment outcomes.

Recently immunological (flowcytometry), and cytogenetic characters namely deletion 17p and immunoglobulin heavy chain gene (IgVH) mutation of CLL patients added more impact of patients' morbidity and response to treatment .

Recent research has focused on the development of targeted therapies for CLL, including venetoclax-based regimens and Bruton tyrosine kinase inhibitors . These agents have shown promise in improving outcomes for patients with CLL, particularly those with high-risk disease or refractory/relapsed disease .

New studies have also explored the role of novel therapies in CLL treatment, including combination regimens and immunotherapies. These approaches have shown encouraging results in early clinical trials, and may offer new options for patients with CLL. in this study we will study the impact of cytogenetics abnormalities [e.g., IGHV mutation status, del(17p)] on patients' treatment response.

A-History taking and clinical examination.

All participants will be subjected to the following: history taking including age at diagnosis, gender, residence, occupation, smoking, comorbidities, duration and symptoms .

Physical findings (lymphadenopathy, splenomegaly, hepatomegaly) Dates of diagnosis, treatment start and type and response to treatment. Treatment and Outcome: First-line therapy, response (CR, PR, SD, PD), follow-up, survival status (PFS, overall survival (OS)) B- Laboratory investigations

Complete blood picture (CBC) with blood film, lymphocytic count Routine liver and kidney function and viral hepatitis Immunophenotyping LDH Coomb's tests Erythrocyte sedimentation rate (ESR). C reactive protein (CRP). Cytogenetic profiles: del(17p) molecular study :IGHV mutation status. C- Other investigation MSCT neck, chest, abdomen, and pelvis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years newly diagnosed with CLL.
* Adequate diagnostics (flowcytometry and cytogenetics) and follow-up data (at least 1 year).
* Patients giving informed consent.

Exclusion Criteria:

* Incomplete diagnostics (e.g. flowcytometry of cytogenetics)
* Lost to follow-up within 12 months of diagnosis.
* Refused to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age ≥ 18 years newly diagnosed with CLL.
  2. Adequate diagnostics (flowcytometry and cytogenetics) and follow-up data (at least 1 year).
  3. Patients giving informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
1)A detailed profile of genetic characteristics in CLL patients . 2)Identification of relation between IGHV Mutation and treatment response.(complete remission,partial remission,stable disease,progressive disease and minimal residual disease response) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mai Mostafa Mohamed, MD, Study Director — assuit univeristy hospitals; Mohamed Ramadan Abdel-Hameed, MD, Study Director — assuit univeristy hospitals

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiorazzi N, Rai KR, Ferrarini M. Chronic lymphocytic leukemia. N Engl J Med. 2005 Feb 24;352(8):804-15. doi: 10.1056/NEJMra041720. No abstract available. PMID 15728813
- [Background] Korsholm C, Bulow C, Christensen M, Dalhoff K, Feinberg JB, Lund TM, Niemann CU, Petersen TS, Andersen MA. Drug exposure and measurable residual disease in chronic lymphocytic leukemia: a systematic review. Leuk Lymphoma. 2025 Feb;66(2):229-239. doi: 10.1080/10428194.2024.2412289. Epub 2024 Nov 7. PMID 39509142